CLINICAL TRIAL: NCT04427982
Title: Dance as an Intervention to Improve Diabetes and Prediabetes Self-Management
Brief Title: Dance and Diabetes/Prediabetes Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00065214
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Diabetes; Pre Diabetes
Keywords: dance; reduce blood sugar; prevention
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: All participants receive the dance and education interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): All participants will attend a 2-month weekly light-to-moderate intensity dance workshop followed by a brief diabetes education and discussion session.
  Interventions: Behavioral: dance; Behavioral: diabetes education

INTERVENTIONS:
Behavioral: dance — Participants will attend a 2-month weekly light-to-moderate intensity dance workshop.
Behavioral: diabetes education — The dance classes will be followed by a brief diabetes education and discussion session.

SUMMARY:
The Dance for Diabetes program was designed as a community service project for the North Carolina Albert Schweitzer Fellowship. The purpose of this research is to evaluate the effectiveness of the project and its impact on participants. This study will assess whether a group dance workshop along with diabetes education can help people with diabetes and prediabetes.

DETAILED DESCRIPTION:
This is a pilot study that will be testing whether or not a group dance workshop is useful and effective. If it is, the study team will refine the workshop model and do additional dance classes in the future. This research study will involve attending a dance workshop once a week for 2 months using an online, video-conferencing computer application. Participants will also receive information about exercise and how to manage their diabetes. Participants will receive a phone call every week during the 2 months to assess their experience. Study participants will also be asked to complete surveys at the beginning and end of the 2-month session, as well as 1 month and 2 months after the classes end.

ELIGIBILITY:
Inclusion Criteria:

* adults proficient in English with diabetes or prediabetes
* subjects who have an established healthcare provider

Exclusion Criteria:

* known cardiovascular disease (acute coronary syndrome, stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack, and peripheral arterial disease) for the last 6 months
* unwilling or unable to partake in light to moderate level of dance physical activity for 1 hour because of physical impairment (e.g. wheelchair, amputation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
National Health and Nutrition Examination Survey Physical Activity and Physical Fitness Questionnaire (NHANES 2019-2020 PAQ)--Activity Confirmation | baseline
  Percentage of subjects who confirm that they are physically active in questionnaire
NHANES 2019-2020 PAQ--Days Active | baseline
  Average number of days subjects report being active
NHANES 2019-2020 PAQ--minutes active | baseline
  Average number of minutes (10-60) per day that participants engage in activity
NHANES 2019-2020 PAQ--Activity Confirmation | 4 weeks post intervention completion
  Percentage of subjects who confirm that they are physically active in questionnaire
NHANES 2019-2020 PAQ--Days Active | 4 weeks post intervention completion
  Average number of days subjects report being active
NHANES 2019-2020 PAQ--minutes active | 4 weeks post intervention completion
  Average number of minutes (10-60) per day that participants engage in activity
NHANES 2019-2020 PAQ--Activity Confirmation | 8 weeks post baseline
  Percentage of subjects who confirm that they are physically active in questionnaire
NHANES 2019-2020 PAQ--Days Active | 8 weeks post baseline
  Average number of days subjects report being active
NHANES 2019-2020 PAQ--minutes active | 8 weeks post baseline
  Average number of minutes (10-60) per day that participants engage in activity
NHANES 2019-2020 PAQ--Activity Confirmation | 8 weeks post intervention completion
  Percentage of subjects who confirm that they are physically active in questionnaire
NHANES 2019-2020 PAQ--Days Active | 8 weeks post intervention completion
  Average number of days subjects report being active
NHANES 2019-2020 PAQ--minutes active | 8 weeks post intervention completion
  Average number of minutes (10-60) per day that participants engage in activity
Diabetes Empowerment Scale (DES) score | baseline
  Score ranges from 1 to 5, with 1 denoting a worse outcome.
DES Score | 4 weeks post intervention completion
  This questionnaire is given to determine if there were any changes in participants' activity level 4 weeks post intervention. Score ranges from 1 to 5, with 1 denoting a worse outcome.
DES score | 8 weeks post baseline
  This questionnaire is given 8 weeks post baseline in order to determine any improvements made during the intervention. Score ranges from 1 to 5, with 1 denoting a worse outcome.
DES Score | 8 weeks post intervention completion
  This questionnaire is given to determine if there were any changes in participants' activity level 8 weeks post intervention. Score ranges from 1 to 5, with 1 denoting a worse outcome.

OTHER OUTCOMES:
Weight | 8 weeks post intervention completion
  measured in kilograms
Body Mass Index (BMI) | 8 weeks post intervention completion
  Weight in kilograms divided by the square of height in meters. A high BMI can be an indicator of high body fatness.
Glycated Hemoglobin (A1c) | 8 weeks post intervention completion
  The A1c test is a blood test that provides information about average levels of blood glucose over the past 3 months. The A1c test can be used to diagnose type 2 diabetes and prediabetes. The A1c test result is reported as a percentage. The higher the percentage, the higher the blood glucose levels have been. A normal A1c level is below 5.7 percent

CONTACTS AND LOCATIONS:
Overall Officials: Julienne Kirk, PharmD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be available immediately following publication without end date.
Access Criteria: Information will be available to anyone who wishes to access the data for any purpose.

DOCUMENTS (1):
  • Informed Consent Form (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT04427982/ICF_000.pdf